CLINICAL TRIAL: NCT02761161
Title: Treatment of Sleep Disturbances in Trauma-affected Refugees: A Randomised Controlled Trial
Brief Title: Treatment of Sleep Disturbances in Trauma-affected Refugees
Acronym: PTF5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Danish Center for Sleep Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PTF5
Record Dates: First submitted 2016-04-27; First posted 2016-05-04 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2017-08

CONDITIONS: Post Traumatic Stress Disorder; Depression
Keywords: PTSD; Sleep; Refugee; IRT; Mianserin
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Mianserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment as usual (No Intervention): TAU: medicine according to algorithm, manual-based cognitive therapy, psychoeducation
- Mianserin (Active Comparator): 10-30 mg of mianserin af sleep enhancing
  Interventions: Drug: Mianserin
- Imagery Rehearsal Therapy (Active Comparator): Therapy focusing on nightmares
  Interventions: Behavioral: Imagery Rehearsal Therapy
- mianserin and Imagery Rehearsal Therapy (Active Comparator): Both mianserin and IRT
  Interventions: Drug: Mianserin; Behavioral: Imagery Rehearsal Therapy

INTERVENTIONS:
Drug: Mianserin — mianserin is add-on treatment to treatment as usual. Max dose 30 mg day.
  Arms: Mianserin; mianserin and Imagery Rehearsal Therapy
Behavioral: Imagery Rehearsal Therapy — IRT is add-on treatment to treatment as usual.
  Other Names: IRT
  Arms: Imagery Rehearsal Therapy; mianserin and Imagery Rehearsal Therapy

SUMMARY:
The overall aim of this study is to examine the effects of sleep enhancing treatment in refugees with PTSD.

DETAILED DESCRIPTION:
BACKGROUND:

Sleep disturbances are often referred to as a hallmark of PTSD. In a sample of 734 trauma-affected refugees undergoing psychiatric treatment at Competence Centre for Transcultural Psychiatry (CTP) in the period 2008-2012 99% reported sleep disturbances and nightmares.

In trauma-affected populations untreated sleep disturbances can uphold and exacerbate both sleep-related and non-sleep-related PTSD symptoms. Sleep disturbances may also affect the efficacy of first-line PTSD treatment and constitute a risk factor for poor outcome of psychiatric treatment. It has been argued that effective treatment of sleep disturbances may accelerate recovery in PTSD. There is a lack of randomised clinical trials on this relation in trauma-affected refugees.

The aim of this study is to examine sleep enhancing treatment in refugees with PTSD.

MATERIALS AND METHOD:

The study will include 230 refugees, diagnosed with PTSD, referred to CTP. Patients who give informed consent will be randomised to four treatment groups.

1. Treatment as usual (TAU); pharmacological treatment according to algorithm and manual based Cognitive Behavioural Therapy
2. TAU and add-on treatment with mianserin
3. TAU and add-on treatment with Imagery Rehearsal Therapy (IRT)
4. TAU and add-on treatment with mianserin and IRT

RESULTS:

This study is expected to bring forward new knowledge on both medical and therapeutic treatment of sleep disturbances in trauma-affected refugees.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Refugees or persons who have been family reunified with a refugee
* PTSD pursuant to the International Classification of Diseases ICD-10 research criteria
* Psychological trauma experienced outside Denmark in the anamnesis. Trauma is imprisonment or detention with torture (according to the United Nation definition of torture) or acts of cruel, inhuman and degrading treatment or punishment. Trauma can also be organised violence, long-term political persecution and harassment, or war and civil war experiences.
* Sleep disturbances/ PSQI >8
* Nightmares/ HTQ score on nightmare item ≥ "a little"
* Signed informed consent

Exclusion Criteria:

* Severe psychotic disorder (defined as patients with an ICD-10 diagnosis F2x and F30.1-F31.9). Patients are excluded only if the psychotic-like experiences are assessed to be part of an independent psychotic disorder and not part of a severe PTSD and/or depression
* Current abuse of drugs or alcohol (F1x.24-F1x.26)
* Known neurodegenerative disorder (Alzheimer's disease (AD), Parkinson's disease (PD), Levy-Body dementia (LBD))
* In need of admission to psychiatric hospital
* Pregnant and breastfeeding women and women of the reproductive age who wish to conceive during the project period.
* Allergy towards active ingredients or excipients in mianserin
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-03; Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Sleep on The Pittsburgh Sleep Quality Index | Change from baseline after approximately 6-8 months treatment

SECONDARY OUTCOMES:
Nightmares on the Disturbing Dreams and Nightmare Severity Index | Change from baseline after approximately 6-8 months treatment
Symptoms of PTSD on The Harvard Trauma Questionnaire | Change from baseline after approximately 6-8 months treatment
Symptoms of depression and anxiety on the Hopkins Symptom Check List | Change from baseline after approximately 6-8 months treatment
Life quality on the WHO-5 | Change from baseline after approximately 6-8 months treatment
level of functioning on the Sheehan Disability Scale | Change from baseline after approximately 6-8 months treatment
Sleep on the REM Sleep Behavior Disorder Screening Questionnaire | 2 years
pain on the Brief Pain Inventory short form | Change from baseline after approximately 6-8 months treatment
Level of functioning on the Global Assessment of functioning - Symptoms | Change from baseline after approximately 6-8 months treatment
Level of functioning on WHODAS 2.0 | Change from baseline after approximately 6-8 months treatment
Symptoms of depression and anxiety on Hamilton depression and anxiety scales | Change from baseline after approximately 6-8 months treatment
Sleep on Actigraph | two weeks recording at baseline and two weeks recording after approximately 6-8 months treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hinuga Sandahl, MD., Principal Investigator — Competence Centre for Transcultural Psychiatry
Locations (1):
- Competence Centre for Transcultural Psychiatry, Copenhagen, Ballerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carlsson J, Bruhn M, Poschmann IS, Silove D, Westergaard ML, Mortensen EL, Sandahl H. Identifying robust predictors of treatment response in trauma-affected refugees: Results from a randomised controlled trial. PLoS One. 2025 Sep 26;20(9):e0324935. doi: 10.1371/journal.pone.0324935. eCollection 2025. PMID 41004514
- [Derived] Sandahl H, Korshoj M, Mortensen OS, Carlsson J. Increase in physical activity is associated with an increase in sleep efficiency, but not with improvement in symptoms of PTSD: analysis of longitudinal data in trauma-affected refugees. J Act Sedentary Sleep Behav. 2024 Feb 15;3(1):7. doi: 10.1186/s44167-024-00046-8. PMID 40217415
- [Derived] Asah C, Sandahl H, Baandrup L, Carlsson J, Jennum P. Dream Enactment Behaviour in Post-Traumatic Stress Disorder. Eur J Psychotraumatol. 2025 Dec;16(1):2444743. doi: 10.1080/20008066.2024.2444743. Epub 2025 Jan 7. PMID 39773112
- [Derived] Sandahl H, Baandrup L, Vindbjerg E, Jennum P, Carlsson J. Social zeitgebers and circadian dysrhythmia are associated with severity of symptoms of PTSD and depression in trauma-affected refugees. Eur Arch Psychiatry Clin Neurosci. 2021 Oct;271(7):1319-1329. doi: 10.1007/s00406-021-01266-8. Epub 2021 May 6. PMID 33956223
- [Derived] Sandahl H, Carlsson J, Sonne C, Mortensen EL, Jennum P, Baandrup L. Investigating the link between subjective sleep quality, symptoms of PTSD, and level of functioning in a sample of trauma-affected refugees. Sleep. 2021 Sep 13;44(9):zsab063. doi: 10.1093/sleep/zsab063. PMID 33710347
- [Derived] Sandahl H, Jennum P, Baandrup L, Poschmann IS, Carlsson J. Treatment of sleep disturbances in trauma-affected refugees: Study protocol for a randomised controlled trial. Trials. 2017 Nov 6;18(1):520. doi: 10.1186/s13063-017-2260-5. PMID 29110681